CLINICAL TRIAL: NCT00953433
Title: Laryngeal Morbidity After Endotracheal Intubation - Endoflex-tube Versus Use of Stylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Martin Kryspin Soerensen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Endoflex-Stylet
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Intubation Complication; Anaesthesia
Keywords: Intratracheal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoflex tube (Experimental): Use of Endoflex tube for intubation.
  Interventions: Device: Endoflex tube
- Endotracheal tube with stylet (Active Comparator): Use of conventional endotracheal tube with a stylet for intubation.
  Interventions: Device: Polyvinyl chloride endotracheal tube with a stylet

INTERVENTIONS:
Device: Endoflex tube — Size decided upon gender.
  Arms: Endoflex tube
Device: Polyvinyl chloride endotracheal tube with a stylet — Size decided upon gender.
  Arms: Endotracheal tube with stylet

SUMMARY:
This study is aimed at reducing the risk of hoarseness and damage to the vocal cords following general anaesthesia. Conventional endotracheal intubation with use of a stylet will be compared with the Endoflex tube. A conventional stylet enforced endotracheal tube is dirigible because of the stiffness gained by the addition of a stylet. In high risk rapid sequence intubation settings the enhanced dirigibility can be crucial, which is why most anaesthesiologists choose to add the stylet in these situations. A new endotracheal tube with a dynamic dirigible end called the Endoflex tube might prove to be a good alternative to the conventional stylet enforced endotracheal tube.

Study hypothesis: The Endoflex tube will reduce the risk of hoarseness after intubation when compared to the conventional stylet enforced endotracheal tube under optimal intubation conditions.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients who require an endotracheal tube during general anaesthesia.
* Informed consent.
* Legally competent.
* Be able to understand Danish and be able to read the given information in Danish.

Exclusion Criteria:

* Planned or former operation in or around the pharynx or the larynx.
* Cancer, infection or sequelae in or around the pharynx or the larynx.
* Use of a stomach tube before or during surgery.
* Suspected difficult intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Postoperative hoarseness | 1 hr postoperatively

SECONDARY OUTCOMES:
Vocal cord sequelae | Preoperative - on average 12 hours before operation
Intubation conditions | During and after intubation - on average 5 minutes
Intubation difficulty scale | During and after intubation - on average 5 minutes
Voice Range Profile | 72 hours postoperatively
  Only for the subgroup of patients with persisting hoarseness
Multi Dimensional Voice Profile | Preoperative - on average 12 hours before operation
Voice Handicap Index | Preoperative - on average 12 hours before operation
Voice Range Profile | After 4 weeks
  Only for the subgroup of patients with persisting hoarseness
Vocal cord sequelae | Within 24 hr postoperatively
Vocal cord sequelae | 72 hours postoperatively
  Only for the subgroup of patients with persisting hoarseness
Vocal cord sequelae | After 4 weeks
  Only for the subgroup of patients with persisting hoarseness
Multi Dimensional Voice Profile | Within 24 hr postoperatively
Multi Dimensional Voice Profile | 72 hours postoperatively
  Only for the subgroup of patients with persisting hoarseness
Multi Dimensional Voice Profile | After 4 weeks
  Only for the subgroup of patients with persisting hoarseness
Voice Handicap Index | After 4 weeks
  Only for the subgroup of patients with persisting hoarseness
Voice Handicap Index | 72 hr postoperatively
  Only for the subgroup of patients with persisting hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rasmussen, MD, PHD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark